CLINICAL TRIAL: NCT06873672
Title: Using EQ-5D-Y to Measure the Health of Patients for Multiple Paediatric Health Conditions: a Project to Validate the Self-complete, Interviewer-administered and Proxy Administered Versions of EQ-5D-Y-3L and EQ-5D-Y-5L in China
Brief Title: Validation of the EQ-5D-Y-3L and EQ-5D-Y-5L for Paediatric Patients in China
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: The EuroQol Research Foundation (Other); Guizhou Provincial People's Hospital (Other); Guizhou Medical University (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Wenjing Zhou, Principal Investigator, RenJi Hospital
Other Study IDs: 2024-IRB-159; 1721-RA (Other Grant/Funding Number: EuroQol Research Foundation)
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Quality of Life (QOL); Patient-Reported Outcome Measures (PROMs); Pneumonia Childhood; Neuroblastoma (NB); Wilms Tumour; Immune Thrombocytopenic Purpura ( ITP )
Keywords: Quality of life; children; psychometric measurements; Paediatric pneumonia; Paediatric central nervous system solid tumour; paediatric immune thrombocytopenic purpura; spillover effect
MeSH Terms: conditions — Neuroblastoma; Wilms Tumor; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Children with pneumonia: Children with pneumonia will be recruited from inpatient wards at Guizhou Provincial People's Hospital and affiliated hospitals of Guizhou Medical University. These children are diagnosed with community-acquired pneumonia (CAP) and receive routine paediatric pneumonia treatment, including antibiotic therapy, oxygen support, intravenous fluids, and symptom monitoring, based on national clinical guidelines.
- Children with central nervous system (CNS) solid tumours: Children with central nervous system (CNS) solid tumours will be recruited from The Children's Hospital affiliated with Zhejiang University School of Medicine. These children are diagnosed with CNS solid tumours, i.e., Neuroblastoma or Wilms tumour, and are either undergoing active treatment (including surgical resection, chemotherapy, and radiotherapy) or in post-treatment follow-up.
- Children with immune thrombocytopenic purpura: Children with immune thrombocytopenic purpura (ITP) will be recruited from paediatric haematology departments at the No.1 Hospital Affiliated to Guizhou Medical University. These children are diagnosed with ITP, a rare autoimmune disorder characterized by low platelet counts and increased bleeding risk. Their treatment varies by disease severity, including observation, corticosteroids, intravenous immunoglobulin (IVIG), or thrombopoietin receptor agonists (TPO-RAs).
- Family caregivers: Caregivers in this study include parents and family caregivers who provide long-term care and support for the child's well-being. Parents (biological or adoptive mothers and fathers) are the primary caregivers, responsible for medical decisions, daily care, and emotional support. Family caregivers, including grandparents, older siblings, aunts, or uncles, may assume caregiving roles due to parental absence or additional support needs, assisting with daily care, medical follow-ups, and emotional well-being.

SUMMARY:
The goal of this observational study is to validate the EQ-5D-Y-3L and EQ-5D-Y-5L in measuring health-related quality of life (HRQoL) for paediatric patients with different health conditions in China. The main research questions focus on comparing the psychometric performance of EQ-5D-Y-3L and EQ-5D-Y-5L, evaluating the differences between self-complete (SC), interviewer-administered (IA), and proxy-administered (Proxy) versions, and assessing their validity against other HRQoL measures like PedsQL. The study will recruit 360 inpatient-caregiver dyads from three disease groups, i.e., pneumonia, paediatric central nervous system (CNS) solid tumours, and immune thrombocytopenic purpura (ITP), using cross-sectional and longitudinal surveys. Baseline assessments will be conducted at hospital admission, with follow-up at hospital discharge (within 14 days). A qualitative component will explore acceptability and interpretation of EQ-5D-Y. The findings will contribute to the methodological development of EQ-5D-Y, with potential implications for HRQoL measurement and economic evaluations in paediatric healthcare.

DETAILED DESCRIPTION:
[Research Background] Health-related quality of life (HRQoL) is a key indicator of well-being in paediatric patients, particularly for those with chronic illnesses. The EQ-5D-Y-3L and EQ-5D-Y-5L are widely used HRQoL measurement tools, but their psychometric properties in Chinese paediatric populations remain underexplored. Understanding how these instruments perform across different administration modes (self-complete, interviewer-administered, and proxy) and in comparison to other established HRQoL measures such as Pediatric Quality of Life Inventory (PedsQL) is essential for improving their application in paediatric healthcare. This study aims to evaluate the validity, reliability, and responsiveness of EQ-5D-Y instruments in children with pneumonia, central nervous system (CNS) solid tumours, and immune thrombocytopenic purpura (ITP) in China, contributing to better HRQoL assessment and economic evaluations in paediatric healthcare.

[Study Design] Prospective observational study.

[Primary Objectives] (1) Compare the psychometric performance (validity, reliability, responsiveness) of EQ-5D-Y-3L and EQ-5D-Y-5L in a Chinese paediatric population. (2) Evaluate differences between self-complete (SC), interviewer-administered (IA), and proxy versions of EQ-5D-Y. (3) Assess how EQ-5D-Y compares with PedsQL in measuring paediatric HRQoL.

[Secondary Objectives] (1) Explore caregiver burden and potential spillover effects using EQ-5D-5L and EQ-HWB-S. (2) Examine the influence of children's disease severity, treatment type, and administration mode on children's HRQoL outcomes. (3) Investigate differences in HRQoL measurement properties across three distinct paediatric disease groups.

[Participants] 360 paediatric patient-caregiver dyads, recruited from three hospitals in China. Disease groups include: Pneumonia (n=120), CNS solid tumours (n=120), and Immune thrombocytopenic purpura (ITP) (n=120).

[Methods] (1) Quantitative assessment: All participants will complete EQ-5D-Y-3L or EQ-5D-Y-5L, administered via three administration modes (SC, IA, or Proxy ). PedsQL will be used as a comparator. Baseline survey will be completed on Day 1 at hospital addmission, and follow-up will occur at discharge (≤14 days) to assess test-retext reliability and responsiveness. (2) Qualitative component: Semi-structured interviews (n=25) will explore acceptability, interpretability, and response patterns.

[Inclusion Criteria] (1) Children aged 5-16 years, diagnosed with pneumonia, CNS solid tumours, or ITP. (2) Primary caregivers (parents/legal guardians) of the participating children. (3) Ability to complete study questionnaires in Mandarin Chinese.

[Study Endpoints] (1) Completion of follow-up assessments. (2) Sufficient qualitative and quantitative data to evaluate HRQoL instruments psychometric properties.

[Primary Outcomes] Psychometric evaluation of EQ-5D-Y, including: Test-retest reliability (intraclass correlation coefficients); Construct validity (correlation with PedsQL, and known-groups validity); Responsiveness (effect size and standardized response means); Comparison of administration modes to determine impact on HRQoL scores.

[Secondary Outcomes] Caregiver burden and spillover Effects will be assessed using EQ-5D-5L and EQ-HWB-S to evaluate caregivers' health and well-being. Correlations with children's HRQoL will explore spillover effects.

[Statistical Methods] (1) Reliability: Test-retest reliability via intraclass correlation coefficients (ICC) and Gwet's AC. (2) Validity: Convergent validity using Spearman's correlation with PedsQL. (3) Known-groups validity assessed via ANOVA and t-tests. (4) Responsiveness: Cohen's d effect sizes and Wilcoxon signed-rank tests. (5) Comparison of administration modes: Generalized linear models (GLM) to assess the impact of SC, IA, and proxy versions on HRQoL scores. (6) Thematic analysis will examine factors contributing to ceiling effects, including response interpretation and differentiation challenges, following COREQ guidelines for rigor. (7) Regression model will be used to analyse the correlation between caregiver's HRQoL and children's.

[Dissemination] This study will provide critical insights into the performance of EQ-5D-Y in China, informing its future use in paediatric health research and economic evaluations. Findings will be disseminated through peer-reviewed publications and international conferences.

ELIGIBILITY:
Inclusion Criteria:

* Children (Patients)

  1. Age: 5-16 years old.
  2. Diagnosis: Clinically confirmed diagnosis of one of the following conditions:

     Pneumonia (hospitalized due to community-acquired pneumonia); Central Nervous System (CNS) Solid Tumours (receiving active treatment or in post-treatment follow-up); Immune Thrombocytopenic Purpura (ITP) (diagnosed with acute or chronic ITP).
  3. Health Status: Cognitively and physically capable of completing HRQoL assessments (for self-complete versions).
  4. Language Proficiency: Able to understand and communicate in Mandarin Chinese.
  5. Consent: Written informed consent obtained from the primary caregiver and verbal or written assent from the child (if age-appropriate).
* Caregivers (Parents/Family Caregivers)

  1. Primary Caregiver: Must be a parent or a long-term family caregiver (e.g., grandparent, older sibling, aunt, or uncle).
  2. Involvement: Directly responsible for the daily care and medical decision-making of the child.
  3. Language Proficiency: Able to understand and complete both the self-complete and proxy-reported HRQoL assessments in Mandarin Chinese.
  4. Consent: Willing to provide informed consent for participation.

Exclusion Criteria:

* Children (Patients)

  1. Severe Cognitive or Developmental Impairment: Diagnosed with intellectual disability, autism spectrum disorder, or any neurological condition that prevents understanding and completing HRQoL assessments.
  2. Severe Physical Disability:

     Conditions that make it impossible to respond to surveys (e.g., advanced neuromuscular disease, severe paralysis).
  3. Comorbidities: Presence of another major chronic illness that could significantly affect HRQoL measurement (e.g., severe congenital heart disease, uncontrolled epilepsy).
  4. Recent Participation in Similar Studies:

     If the child has participated in another HRQoL validation study within the past 6 months.
  5. Inability to Complete Study Follow-Up: Expected to be transferred to another hospital or relocated during follow-up.
* Caregivers (Parents/Family Caregivers)

  1. Not the Primary Caregiver:
  2. Individuals who do not have daily caregiving responsibilities for the child.

     Cognitive Impairment or Severe Health Conditions:
  3. Caregivers with severe mental illness, dementia, or a medical condition that affects their ability to complete surveys.
  4. Language Barrier: Unable to understand and complete HRQoL assessments in Mandarin Chinese.
  5. Refusal to Participate: Caregivers who decline to provide informed consent.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited from three tertiary hospitals different cities in China.
  The study will enroll paediatric patients aged 5-16 years who are receiving routine care for pneumonia, central nervous system (CNS) solid tumours, or immune thrombocytopenic purpura (ITP). These conditions represent common and clinically significant paediatric health issues requiring hospitalization or specialized treatment.
  The study will also recruit primary caregivers, who are typically parents or long-term family caregivers responsible for the child's daily care and medical decision-making.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in EQ-5D-Y Summary Scores across three disease groups from Baseline to Follow-up | From Day 1 (hospital admission) to hospital discharge (within 14 days)
  The EQ-5D-Y Summary Scores include: (1) Index Score which is derived using the Chinese value set for EQ-5D-Y-3L; (2) the Level Sum Score (LSS) which is calculated by summing the reported levels across five dimensions of the EQ-5D-Y-3L and EQ-5D-Y-5L (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), with higher scores indicating worse health; and (3) the visual analogue scale (EQ VAS), a self-reported global health assessment measured on a 0 to 100 scale, where 0 represents the worst imaginable health and 100 represents the best imaginable health. The change in these scores from baseline to follow-up will be analyzed to assess test-retest reliability, responsiveness and known-groups validity, and will be compared across the three administration modes (self-complete, interviewer-administered, and proxy-reported) and across three disease groups.

SECONDARY OUTCOMES:
Caregiver Burden and Spillover Effects Using EQ-5D-5L and EQ-HWB-S | At hospital admission (Day 1)
  The impact of caregiving burden on parents will be assessed using the EQ-5D-5L and EQ Health and Well-Being Scale (EQ-HWB-S), both of which generate preference-based index scores. The EQ-5D-5L assesses caregivers' health status across five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-while the EQ-HWB-S captures a broader range of well-being aspects, including social and emotional impacts such as exhaustion, loneliness, and cognitive difficulties. Index scores for both instruments will be derived using the respective value sets, with higher scores indicating better health and well-being. Correlations between caregiver scores and children's EQ-5D-Y scores will be analyzed to explore spillover effects, distinguishing between caregiving-related burdens and broader family-level impacts.

CONTACTS AND LOCATIONS:
Locations (1):
- Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Qi X, Zhou W, Yang Z, Guannan B, Yang X, Zhang J, Busschbach J. Validation of EuroQol instruments in paediatric patients and their caregivers in China: protocol for a prospective observational study. BMJ Open. 2025 Jun 18;15(6):e102509. doi: 10.1136/bmjopen-2025-102509. PMID 40533211